CLINICAL TRIAL: NCT01285050
Title: Interferon Alfa Sensitivity in HIV/HCV Coinfected Persons Before and After Antiretroviral Therapy
Brief Title: Interferon Alfa Sensitivity in HIV/HCV Persons Before and After HIV Meds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, David Thomas, Chief, Infectious Diseases, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NA00040361; R01DA013806 (NIH)
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: HIV Infection; Hepatitis C
Keywords: HIV; Human immunodeficiency virus; Acquired Immune Deficiency Syndrome Virus; AIDS Virus; Immunodeficiency Virus, Human; Virus, Human Immunodeficiency; Hepatitis C; Hepatitis C, chronic; Hepatitis C virus; Hepatitis C antibodies; Hepatitis C antigens
MeSH Terms: conditions — HIV Infections; Hepatitis C; Acquired Immunodeficiency Syndrome; Hepatitis C, Chronic | interventions — Antiretroviral Therapy, Highly Active; Raltegravir Potassium; Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pre post ART (Other): HCV and HIV viral load pre and post antiretroviral therapy (ART). ART is the intervention and the comparison is the HIV and HCV viral load reductions as determined by RT-PCR after administration of interferon alfa in each instance (before and after ART)
  Interventions: Drug: Antiretroviral therapy (ART); Drug: raltegravir; Drug: Emtricitabine and tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Antiretroviral therapy (ART) — Peginterferon alfa-2b administered once as part of a pharmacokinetic study before and after anti-HIV medications. Peginterferon is used to produce a measurement but the intervention is the HIV medications which are specified as raltegravir, emtricitabline, and tenofovir disoproxil fumerate.
Drug: raltegravir — raltegravir is an HIV medication given 400 mg twice daily by mouth
  Other Names: Isentress
Drug: Emtricitabine and tenofovir disoproxil fumarate — Emtricitabine and tenofovir disoproxil fumarate are HIV medications, combination pill, once per day by mouth
  Other Names: Truvada

SUMMARY:
The chief purpose of this research is to evaluate interferon alpha sensitivity and cell type specific levels of interferon receptor and interferon stimulated genes and proteins in HIV/ HCV (hepatitis C virus) coinfected persons before and after administration of HIV medications (antiretroviral therapy).

DETAILED DESCRIPTION:
We plan to perform liver biopsy by microlaparoscopy on previously untreated HIV/HCV coinfected persons, then give them a dose of peginterferon alfa 2b. HCV and HIV kinetics will be studied. Afterward, HIV will be treated using antiretroviral therapy and the procedure will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Adult Human
* Able to provide written informed consent
* HIV antibody positive
* HIV viral load positive
* HIV treatment naive
* Hepatitis C antibody positive
* Hepatitis C viral load positive
* Hepatitis C treatment naive
* Approved to take HIV medications for minimum 9 months
* Willing to use contraception, Life expectancy greater than 2 years

Exclusion Criteria:

* Significant opportunistic infections within 12 month
* Hepatitis B positive
* Evidence of liver cirrhosis
* Decompensated liver disease
* Chronic alcohol abuse
* Allergy to raltegravir, tenofovir, and/or emtricitabine
* Active or suspected malignancy
* Sarcoidosis
* Active TB
* Coronary artery disease
* Uncontrolled seizures
* Untreated thyroid disease
* Untreated diabetes
* Weight greater than 125 kg
* Severe depression or severe psychiatric disorder
* Ongoing alcohol or illicit drug use
* Pregnant, nursing, pr planning to become pregnant
* Allergy to interferon

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Kandathil AJ, Breitwieser FP, Sachithanandham J, Robinson M, Mehta SH, Timp W, Salzberg SL, Thomas DL, Balagopal A. Presence of Human Hepegivirus-1 in a Cohort of People Who Inject Drugs. Ann Intern Med. 2017 Jul 4;167(1):1-7. doi: 10.7326/M17-0085. Epub 2017 Jun 6. PMID 28586923
- [Derived] El-Diwany R, Breitwieser FP, Soliman M, Skaist AM, Srikrishna G, Blankson JN, Ray SC, Wheelan SJ, Thomas DL, Balagopal A. Intracellular HIV-1 RNA and CD4+ T-cell activation in patients starting antiretrovirals. AIDS. 2017 Jun 19;31(10):1405-1414. doi: 10.1097/QAD.0000000000001480. PMID 28358734

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre Post ART: HCV and HIV viral load pre and post antiretroviral therapy
  Anti-HIV Agents: Interferon alfa-2b administered once as part of a pharmacokinetic study before and after anti-HIV medications.
  raltegravir: HIV medication, 400 mg twice daily by mouth
  Emtricitabine and tenofovir disoproxil fumarate: HIV medication, combination pill, once per day by mouth
Period: Overall Study
Arm/Group | Pre Post ART
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pre Post ART
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
HCV infected [Number; unit: participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: HCV RNA
Description: HCV RNA determined by reverse transcription polymerase chain reaction and measured as log IU/ml 48 hours after a single dose of peginterferon alfa 2b 1.5 μg/kg.
Time Frame: 48 hours after interferon administration
Measure: Median (Inter-Quartile Range); unit: log IU/ml
Groups:
- Pre ART HCV RNA Decline: HCV viral load determined by RT-PCR and reported as log IU/ml before giving antiretroviral therapy (ART)
  Interferon alfa-2b was administered once as part of a pharmacokinetic study before and after ART.
  ART included:
  raltegravir: HIV medication, 400 mg twice daily by mouth
  Emtricitabine and tenofovir disoproxil fumarate: HIV medication, combination pill, once per day by mouth
- Post ART HCV Decline: HCV RNA determined by RT-PCR and expressed as log IU/ml after ART
Arm/Group | Pre ART HCV RNA Decline | Post ART HCV Decline
Number analyzed (Participants) | 19 | 19
log IU/ml | 0.65 [0.17 to 1.15] | 0.81 [0.34 to 1.47]

ADVERSE EVENTS:
Arm/Group | Pre Post ART
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre Post ART (N=20)
bleeding (Injury, poisoning and procedural complications) | 1 (1) — As an expected potential complication of liver biopsy, one patient had bleeding that required observation in the hospital. No residual complications were noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No